CLINICAL TRIAL: NCT00263081
Title: A Double-blind, Placebo-controlled, Randomized Study to Evaluate the Efficacy and Safety of TAK-475 or Placebo When Co-administered With Current Lipid-lowering Therapy in Subjects With Homozygous Familial Hypercholesterolemia.
Brief Title: Efficacy of Lapaquistat Acetate Co-Administered With Current Lipid-Lowering Treatment on Blood Cholesterol Levels in Subjects With Homozygous Familial Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Overall profile of the compound does not offer significant clinical advantage to patients over currently available lipid lowering agents
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-475-016; 2005-003626-26 (EudraCT Number); U1111-1122-7919 (Registry Identifier: WHO)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate QD (Experimental): (and current lipid-lowering treatment)
  Interventions: Drug: Lapaquistat acetate and current lipid-lowering treatment
- Current lipid-lowering treatment (Placebo Comparator)
  Interventions: Drug: Current lipid-lowering treatment

INTERVENTIONS:
Drug: Lapaquistat acetate and current lipid-lowering treatment — Cohort 1: Weight is less than 50 kg:
  Lapaquistat acetate 50 mg, tablets, orally, once daily and current lipid-lowering treatment for up to 12 weeks.
  Cohort 2: Weight is more than 50 kg:
  Lapaquistat acetate 100 mg, tablets, orally, once daily and current lipid-lowering treatment for up to 12 weeks.
  Other Names: Lapaquistat; TAK-475
  Arms: Lapaquistat Acetate QD
Drug: Current lipid-lowering treatment — Lapaquistat acetate placebo-matching tablets, orally, once daily and current lipid-lowering treatment for up to 12 weeks.
  Arms: Current lipid-lowering treatment

SUMMARY:
The purpose of the study is to determine the efficacy of lapaquistat acetate, once daily (QD), to lower cholesterol in subjects with homozygous familial hypercholesterolemia undergoing lipid-lowering treatment.

DETAILED DESCRIPTION:
According to the World Health Organization, CHD is now the leading cause of death worldwide. In 2001, CHD caused 7.2 million deaths and estimates for 2020 indicate that annual CHD deaths will increase to 11.1 million. These statistics suggest that improved options are needed to treat hypercholesterolemia and dyslipidemia.

The balance among cholesterol synthesis, dietary intake, and degradation is normally adequate to maintain healthy cholesterol plasma levels. However, in patients with hypercholesterolemia, elevated low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls. Consequently, in this population it has been established that lowering low-density lipoprotein cholesterol plasma concentrations effectively reduces cardiovascular morbidity and mortality. The National Cholesterol Education Program Adult Treatment Panel III has therefore identified control of low-density lipoprotein cholesterol as essential in the prevention and management of CHD. Additional lipid risk factors designated by National Cholesterol Education Program Adult Treatment Panel III include elevated triglycerides, elevated non-high-density lipoprotein cholesterol (atherogenic lipoproteins), and low levels of high-density lipoprotein cholesterol. Lipoproteins rich in triglycerides, such as very-low-density lipoprotein cholesterol, appear to contribute to atherosclerosis, whereas the apparent protective effect of high-density lipoprotein cholesterol, which is likely related to high-density lipoprotein cholesterol-facilitated transport of cholesterol away from atherosclerotic deposits, may be limited at low high-density lipoprotein cholesterol concentrations.

Initial dietary and lifestyle measures taken to control dyslipidemia are often inadequate, and most patients require pharmacologic intervention. Currently, 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (statins) are the first-line monotherapies most often prescribed to reduce low-density lipoprotein cholesterol, after diet and therapeutic lifestyle change. However, with statin monotherapy, many patients fail to reach National Cholesterol Education Program Adult Treatment Panel III recommended levels of low-density lipoprotein cholesterol reduction. As a result, the statin dosage must be increased or an additional treatment added to achieve treatment goals. Increasing the statin dosage may result in decreased tolerability and potential safety concerns, contributing to the high discontinuation rates of statins and their prescription at low and often ineffective doses. Further, although the effectiveness of increasing the dose varies among the statins, in general, doubling of the dose above the minimum effective dose has been found to decrease serum low-density lipoprotein cholesterol by only an additional 6 percent.

Takeda Global Research and Development Center, Inc. is developing an orally active squalene synthase inhibitor, TAK-475 (lapaquistat acetate) for the treatment of dyslipidemia. Lapaquistat acetate inhibits the biosynthesis of cholesterol by inhibiting the enzyme squalene synthase, which catalyzes the conversion of farnesyl diphosphate to squalene-a precursor in the final steps of cholesterol production.

This study will evaluate the efficacy of lapaquistat acetate coadministered with ongoing lipid-lowering therapy in treating subjects with homozygous familial hypercholesterolemia. The effect on LDL-C and other lipid parameters, as well as the safety and tolerability of lapaquistat acetate compared to a placebo will be evaluated during a 12-week double-blind treatment period. The long-term safety of lapaquistat acetate treatment in this population will be evaluated during an open-label extension period. Study Participation is anticipated to be up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 8 years of age (12 years of age in Poland) and weigh greater than or equal to 30 kg.
* Must have homozygous FH, as documented by genetic testing that confirmed 2 mutated alleles at the LDL-receptor locus, or by the following clinical criteria:

  * documented history of untreated fasting serum LDL-C >460 mg/dL (11.91 mmol/L).
  * tendinous or cutaneous xanthomas and/or corneal arcus before age 10 and/or premature coronary heart disease before age 20.
* Must be taking a stable, approved lipid-lowering drug regimen for a minimum of 8 weeks prior to Screening Visit 1 and were to continue that treatment for the duration of the study.
* Female participants can not be pregnant, not lactating, not planning on becoming pregnant and agree to use adequate contraception throughout the course of the study.

Exclusion Criteria:

* Has alanine aminotransferase or aspartate aminotransferase levels greater than 2 times the upper limit of normal, active liver disease, jaundice, or serum creatinine >135 μmol/L (1.5 mg/dL) at screening.
* Has a creatine kinase greater than 3 times the upper limit of normal
* Has a positive hepatitis B surface antigen, or hepatitis C virus antibody, as determined by medical history.
* Has a positive human immunodeficiency virus status or was taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Is unable or unwilling to discontinue excluded medications or to continue stable doses of 'stable dose' medications or would require treatment with any excluded medication during the study.
* Is currently participating in another investigational study or had participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study drug. This criterion was not to include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.
* Has known hypersensitivity or history of adverse reaction to lapaquistat acetate.
* Has a history of fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has an endocrine disorder, such as Cushing Syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism. Subjects with hypothyroidism on appropriate replacement therapy.
* Has uncontrolled hypertension despite medical treatment.
* Has inflammatory bowel disease or any other malabsorption syndrome or had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Has any other serious disease or condition at screening or at randomization that might have reduced life expectancy, impaired successful management according to the protocol, or made the subject an unsuitable candidate to receive study drug.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Low Density Lipoprotein cholesterol | Week 12 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in calculated Low Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Triglycerides | Week 12 or Final Visit
Change from Baseline in Total Cholesterol | Week 12 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 12 or Final Visit
Change from Baseline in apolipoprotein B | Week 12 or Final Visit
Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 12 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (10):
- United States (2):
  - Cincinnati, Ohio
  - Columbus, Ohio
- Québec, Canada
- France (2):
  - Paris
  - Strasbourg
- Jerusalem, Israel
- Poland (3):
  - Bialystok
  - Warsaw
  - Zabrze
- Manchester, United Kingdom

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985